CLINICAL TRIAL: NCT03548844
Title: A Prospective Randomized Controlled Trial Of Local Excision Versus Total Mesorectal Excision In Pathological Complete Response (ypT0-1cN0) Mid- or Low-Rectal Cancer After Neoadjuvant Therapy
Brief Title: Local Excision Versus Total Mesorectal Excision In Pathological Complete Response (ypT0-1cN0) Mid- Or Low-Rectal Cancer After Neoadjuvant Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, MD,PhD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRSSYSU01
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Rectal Cancer; Surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: This trial is a a two-arm, open labelled, prospective, randomized phase III studies. Eligible patients with ypT0-1cN0 rectal cancer patients will be randomly assigned, in a 1:1 ratio, to receive either observation (local excision group) or complementary rectal excision (total mesorectal excision group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local excision group (Experimental): Pathologically verified ypT0-1cN0 rectal cancer patients after local excision are randomized to observation (local excision group)
  Interventions: Procedure: local excision
- total mesorectal excision group (Active Comparator): Pathologically verified ypT0-1cN0 rectal cancer patients after local excision are randomized to complementary rectal excision (local excision group)
  Interventions: Procedure: total mesorectal excision

INTERVENTIONS:
Procedure: local excision — Pathologically verified ypT0-1cN0 rectal cancer patients after local excision are randomized to observation (local excision group) .
  Arms: local excision group
Procedure: total mesorectal excision — Pathologically verified ypT0-1cN0 rectal cancer patients after local excision are randomized to complementary rectal excision (total mesorectal excision group).
  Arms: total mesorectal excision group

SUMMARY:
Patients with cT2-4aN0-2M0 mid- or low-rectal cancer received neoadjuvant chemotherapy or combined chemoradiotherapy. Good responders (cT0-1N0) patients received local excision 4-8 weeks after treatment. Pathologically verified ypT0-1 patients are randomized to observation (local excision group) or complementary rectal excision (total mesorectal excision group). The composite end points include 3 year disease-free survival (DFS), overall survival (OS), recurrence, major morbidity and quality of life.

DETAILED DESCRIPTION:
Total mesorectal excision is still the standard surgical treatment of mid-and low advanced rectal cancer after neoadjuvant treatment. This radical procedure inevitably has the risk of major short and long term morbidity and anorectal function impairment. Additionally, abdominal perineal resection(APR) with permanent stoma is still applied to some low rectal cancer patients, even though major response had been achieved after neoadjuvant treatment. Previous studies have proposed "wait and see" strategy in clinical complete response patients. The local recurrence rate is still high due to residue adenocarcinoma lesion.

Local excision is a conservative alternative approach associated with low mortality and morbidity and high quality of life. In this study, the investigators proposed local excision in good responders (cT0-1N0) 4-8 weeks after neoadjuvant treatment. Patients with pathologically verified complete response (ypT0-1cN0) are randomized to observation (local excision group) or complementary rectal excision (total mesorectal excision group). The purpose of this prospective randomized controlled study is to compare local excision versus total mesorectal excision in pathological complete response (ypT0-1cN0) mid- or low-rectal cancer after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1、Willing and able to provide written informed consent. 2、Histological or cytological documentation of adenocarcinoma of the rectum (≤8 cm from the anal verge).

  3、ypT0-1cN0 after neoadjuvant therapy 4、No metastatic disease. 5、Patient is at least 18 years of age. 6、Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 7、Non complicated primary tumor (obstruction, perforation, bleeding).

Exclusion Criteria:

* 1、T1, T4 tumour or anal sphincter invasion 2、Metastatic disease (M1) 3、Contra indication for radiotherapy and/or fluoropyrimidine use in chemotherapy 4、Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study 5、History of cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
DFS | 3 years
  Disease-free survival

SECONDARY OUTCOMES:
OS | 3 years
  Overall survival
Morbidity rate | 1 year
  Morbidity rate
Mortality rate | 1 year
  Mortality rate
Anorectal function outcomes | 3 years
  To evaluate defecating function with Wexner score
Quality of life | 3 years
  To evaluate quality of life with EORTC QLQ-30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Liang Kang, MD,PhD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China